CLINICAL TRIAL: NCT05918653
Title: Demographic, Clinical, and Biomedical Profile of Diabetic Patients Receiving Home Healthcare in Saudi Arabia
Status: Completed | Type: Observational
Sponsor: Saudi Scientific Home Health Care Society (Other)
Responsible Party: Principal Investigator, Lamya Mohammed Alzubaidi, Principal Investigator, Saudi Scientific Home Health Care Society
Other Study IDs: 01
Record Dates: First submitted 2023-06-14; First posted 2023-06-26 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Home Healthcare — No intervention in this study
  Other Names: No intervention in this study

SUMMARY:
Background: Identifying characteristics of diabetic patients receiving home healthcare will help in designing services that respond to their conditions and improve their health status and quality of life. The aim of this study is to describe demographic, clinical, and biomedical characteristics of diabetic patients receiving home healthcare.

Methodology:

Descriptive cross-sectional study was conducted in King Salman Hospital in Riyadh, and Al Madinah home healthcare center in Saudi Arabia. The study Population included diabetic patients receiving home healthcare from these two health institutions. The inclusion criteria were type 1 and type 2 diabetes mellitus, all age groups, both males and females. A sample of 239 diabetic patients was selected using the stratified random sampling technique. Data were collected from the medical records of the eligible, selected study population using a structured data collection sheet. Data were analysed by statistical Package for the Social Sciences (SPSS) version 21. Categorical data were expressed as percentages with 95% confidence intervals, continuous data as mean and standard deviations.

DETAILED DESCRIPTION:
Background:

Diabetes Mellitus (DM) is a chronic disease that affects approximately 194 million individuals, equivalent to 5.1% of the adult population globally1. In Saudi Arabia, the age-adjusted prevalence of diabetes is currently estimated to be 18.7% according to the International Diabetes Federation2. This high prevalence places the country among the top five in the Middle East and North Africa region 2 and top ten globally3.

DM can cause acute medical crises, such as diabetic ketoacidosis4, as well as long-term complications, including blindness, renal failure, and lower limb amputations1. These complications can cause significant suffering for individuals and have a considerable impact on their quality of life and overall health outcomes1,4.

To effectively prevent medical crises and long-term complications associated with diabetes, access to ongoing and timely care is crucial, and flexible follow-up schedules must also be in place to ensure comprehensive management of the disease4,5. However, the access and scheduling limitations associated with traditional clinic-based medical care might hinder the provision of such care5. Consequently, home-based care has emerged as a convenient alternative for the provision of diabetes management, particularly for elderly individuals and patients who are house-bound or bed-dependent.

Home healthcare (HHC) is a recognized model of healthcare provision that encompasses a broad range of medical and health services delivered by skilled practitioners in the patient's home6-7. DM is currently located behind congestive heart failure as the primary diagnosis for admission to HHC7,8. In Saudi Arabia, patients with diabetes mellitus are among the seventeen categories that qualify for HHC services provided by the Ministry of Health(MoH)9.

Numerous studies have evaluated the characteristics of diabetic patients in Saudi Arabia, including their glycaemic control levels3,10,11. However, there is a lack of data regarding diabetic patients who receive HHC. These patients may differ from the general diabetic population, as they may be older and experience mobility restrictions due to underlying conditions. Consequently, there is a pressing need to identify the profile of these patients to determine their current situation and to inform the development of tailored HHC services that enhance their health outcomes and overall quality of life.

1. Objective:

2.1. General Objective To assess the Current situation of diabetic patients receiving Home Health Care in Riyadh and Medina Regions 2.2. Specific Objectives:

1. To identify the characteristics of diabetic patients receiving Home Health Care in Riyadh and Medina Regions with regards to:

   * General background
   * Medical and biomedical
   * Use of outpatient services
   * Admission to hospital
2. To describe the home healthcare provided to diabetic patients in Riyadh and Medina Regions with regards to:

   * Types of services
   * Type of home healthcare provider

2. Material and methods: 2.3. Study design: Descriptive cross-sectional study 2.4. Study area: 3. Study was conducted in the King Salman Hospital and Al Madinah Home Healthcare center. King Salman hospital was the first hospital to start the provision of homecare services in Riyadh region in 2005. Currently the hospital has 390 patients receiving home healthcare, around 50% of them have DM. Al Madinah Home Healthcare center was also established in 2005 and currently provides care to 581 patients, with approximately 86% of them diagnosed with DM. The scope of the services provided under the home healthcare in both centers covers diagnosis, management and follow-up of patients. Both HHC centers belong to the Saudi MoH and provide HHC services according to the regulations of the General Directorate of HHC in the MoH.

3.1. Study population: Diabetic patients receiving home healthcare by King Salman Hospital and Al Madinah Home healthcare center.

o Inclusion criteria:

* Type1 and type 2 diabetes mellitus
* All age groups
* Males and females 3.2. Sampling: • Sampling technique: The sample was selected using the stratified random sampling technique. The calculated sample size was divided between the King Salman homecare centre and Al Madinah homecare centre according to the weight of diabetic patients in each centre. From each centre the diabetic patients were selected using the simple random sampling technique.

  * Sample size:

Population size(for finite population correction factor or fpc)(N): 630 Hypothesized % frequency of outcome factor in the population (p): 50%+/-5 Confidence limits as % of 100(absolute +/- %)(d): 5% Confidence level 95%

The sample was calculated using the calculator of the Open Source Statistics for Public Health [13] assuming the following inputs:

This this yielded a sample size of 239 diabetic patients.

3.3. Data collection technique and tool: 3.3.1. Source of data:

* Medical records of diabetic patients receiving home health care from King Salman hospital in Riyadh and Al Madinah Home healthcare center in Al Madinah.
* Data were collected a structured, per-coded data collection sheet composed of the following sections:

  * General background information:

    * Sociodemographic characteristics (age, gender…. etc.)
    * Presence of care giver
    * Knowledge of caregiver
  * Medical information:

    * Type of diabetes
    * Medication
    * Duration of diabetes
    * Co-morbidities
    * Diabetes complications
    * Admission to hospital
    * Use of outpatient services
  * Biomedical information:

    * Blood pressure
    * Weight, height (BMI)
    * Glycated hemoglobin.
    * Fasting blood glucose (FBG),
    * Serum creatinine
  * Home healthcare

    * The types of homecare health services received
    * Type of healthcare professional providing the home healthcare
    * The frequency of the home healthcare per week/month
    * The duration of the home healthcare 3.4. Data analysis plan: Data entry and analysis were performed using Statistical Package for the Social Sciences software version 21. The data were summarized and presented as frequencies and percentages for categorical data, and means (± standard deviation) for normally distributed numerical data, and medians (range) for skewed numerical data. Using the HbA1c values, the study population was divided into two categories (HbA1c <8% and HBA1c ≥8%) according to The Saudi National Diabetes Center (SNDC) guidelines for elderly diabetic patients with comorbidities. The eGFR was calculated using age, sex, ethnicity and creatinine level, and the population was grouped based on SNDC guidelines as eGFR <60 or ≥60 mL/min/1.73m2.

3.5. Ethical considerations: The research was considered exempt from review by the Institutional Review Board (IRB) of Prince Nourah bint Abdulrahman University ( IRB log number:22-1051).

ELIGIBILITY:
Inclusion Criteria:

* Type1 and type 2 diabetes mellitus
* All age groups
* Males and females
* Receiving home healthcare

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with diabetes milletus receiving home healthcare from King Salman Hospital in Riyadh and Al Madinah Home healthcare center in Al Madinah, Saudi Arabia
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Biomedical profile of diabetic patients | three months
  proportion of diabetic patients with Glycated haemoglobin less than 8%

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Al Madinah Home Healthcare center, Al Madīnah
  - King Salman Hospital, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Diabetes Federation. (2003). Diabetes Atlas (2nd ed.). Brussels, Belgium: International Diabetes Federation
- [Background] International Diabetes Federation.(2021). Diabetes in Middle-East & North Africa
- [Background] Alshareef SM, Aldayel AY, AlKhathlan MA, Alduaij KO, Alshareef FG, Al-Harthi ME, Aldayel AA, Shadid AM, Dahmash AB. Diabetic patients in Saudi Arabia: The evaluation of glycemic control measures based on emergency department utilization and the percentages of adherence to the recommended follow-ups for microvascular complications. Saudi Med J. 2019 Mar;40(3):271-276. doi: 10.15537/smj.2019.3.23968. PMID 30834423
- [Background] Kitabchi AE, Umpierrez GE, Miles JM, Fisher JN. Hyperglycemic crises in adult patients with diabetes. Diabetes Care. 2009 Jul;32(7):1335-43. doi: 10.2337/dc09-9032. No abstract available. PMID 19564476
- [Background] Hartman A, Creek W, Care H. In-Home Chronic Disease Management in Diabetes A Collaborative Practice Model for Home. Home Health Care Management & Practices
- [Background] Almoajel A, Al-Salem A. The Quality of Home Healthcare Service in Riyadh/Saudi Arabia. AjscLeena-LunaCoJp
- [Background] Sertbas M, Guduk O, Guduk O, Yazici Z, Dagci S, Sertbas Y. Current situation analysis of diabetic home care patients. North Clin Istanb. 2019 Oct 25;7(2):140-145. doi: 10.14744/nci.2019.59751. eCollection 2020. PMID 32259035
- [Background] O'Reilly CA. Managing the care of patients with diabetes in the home care setting. Diabetes Spectr
- [Background] Depuityship of theraputic care. home healthcare manual. Ministry of Health. Riyadh Saudi Arabia
- [Background] Alramadan MJ, Magliano DJ, Almigbal TH, Batais MA, Afroz A, Alramadhan HJ, Mahfoud WF, Alragas AM, Billah B. Glycaemic control for people with type 2 diabetes in Saudi Arabia - an urgent need for a review of management plan. BMC Endocr Disord. 2018 Sep 10;18(1):62. doi: 10.1186/s12902-018-0292-9. PMID 30200959
- [Background] Elhadd TA, Al-Amoudi AA, Alzahrani AS. Epidemiology, clinical and complications profile of diabetes in Saudi Arabia: a review. Ann Saudi Med. 2007 Jul-Aug;27(4):241-50. doi: 10.5144/0256-4947.2007.241. PMID 17684435